CLINICAL TRIAL: NCT05464524
Title: The Role of Various Environmental Factors on the Incidence, Severity and Recurrence of Diabetic Foot Ulcers (DFUs) in Adult Patients With Diabetes in England
Brief Title: Environmental Factors on DFUs Incidence - a Mixed-mode Survey
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Biotherapy Services Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: 312284
Record Dates: First submitted 2022-07-04; First posted 2022-07-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer
Keywords: diabetic foot ulcer; diabetes; environmental factors
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Main questionnaire — 10-15 minute questionnaire asking about environmental factors (i.e daily lifestyle questions), quality of life, comorbidities among others.
Other: Optional 12-week follow up questionnaire — A 5-minute questionnaire asking about changes to the quality of life and DFU status since the initial questionnaire.

SUMMARY:
Diabetic foot ulcers (DFUs) pose a significant threat to the health and wellbeing of diabetic patients. Affecting around 1 in 10 people (NHS North West Coast Strategic Clinical Networks, 2017) regardless of a diabetes type they often result in a drastically worsened quality of life and can lead to severe consequences including leg amputations. This survey will help to understand what role various environmental factors have on the incidence, severity and recurrence of DFUs. Results from this study will help healthcare professionals as well as patients to better understand various factors involved in DFU prevalence. Moreover, this survey could help to appreciate whether a more holistic approach should be followed when assessing DFU risk and deciding on therapy. This study will be run across five sites in England between October 2023 and May 2024 and will involve a small pilot study (informal interview) and an anonymous, ten-minute questionnaire. Any adult with an ongoing or past DFU will be eligible. Participants will be asked about their job type, quality of life, diabetic therapy, comorbidities, and environmental factors questions. There will be an option for a follow-up questionnaire after 12 weeks to understand the healing process and changes to the quality of life following a DFU incident. Additionally, patients may consent to provide access to excerpts from their anonymized medical history details (prescribed medications) to better understand their diabetic and DFU history. This study will be run as part of an industrial, London Interdisciplinary Biosciences Consortium (LIDo) PhD project investigating the autologous platelet-rich plasma gel for diabetic foot ulcers (RAPID™ biodynamic haematogel) with King's College London as funded by the Biotechnology and Biological Sciences Research Council (BBSCR) and Biotherapy Services Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (>18 years old)
2. Diagnosed with diabetes
3. Currently having or have had at least one diabetic foot ulcer incident in the past
4. Resident in England
5. Able to consent

Exclusion Criteria:

1. Underaged
2. Not diagnosed with diabetes
3. Never had a DFU incident
4. Unable/refusing to consent
5. A non-English resident

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult English residents with a past or present diabetic foot ulcer.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Established the role of tested environmental factors and lifestyle choices on the incidence, recurrence, and severity of diabetic foot ulcers in adults living with diabetes in England. | 9 months
  Descriptive statistics used to characterise the study population. Logistic regression modelling of tested environmental factors to establish models quantifying the association between independent and dependent variables (DFU incidence, severity, recurrence).
  Identified main environmental factors that produce the highest probability of having a severe diabetic foot ulcer case (based on the answers to the EQ-5D-5L - a severe DFU incident would is predicted to influence mobility, self-care, pain levels, performance of usual activities and anxiety/depression.)

SECONDARY OUTCOMES:
Quantified the associations between the other disease co-occurring with diabetes and the medications or therapies prescribed for them that may have an impact on diabetic foot ulcer incidence and severity. | 9 months
  - Logistic regression models obtained to understand the association between diabetic comorbidities/prescribed medications and the characteristics of a diabetic foot ulcer (severity and recurrence).
Established changes to DFU status and quality of life over the 12 week follow up period. | 9 months
  Quantified the change in quality of life over 12-week period and testing the association by performing a t-test between the DFU incident outcome and quality of life (based on the answers to the EQ-5D-5L).

CONTACTS AND LOCATIONS:
Overall Officials: Ben Forbes, Professor, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only processed data will be shared. No individual responses/raw data is planned to be shared with other researchers.